CLINICAL TRIAL: NCT02548494
Title: Early Administration of Long-acting Insulin Glargine for the Treatment of Diabetic Ketoacidosis in Pediatric Type 1 Diabetes: A Randomized Double Blind Trial
Brief Title: Early Administration of Long-acting Insulin Treatment of Diabetic Ketoacidosis in Pediatric Type 1 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Project terminated due to insufficient resources for recruitment.
Sponsor: Chattanooga-Hamilton County Hospital Authority (Other)
Responsible Party: Principal Investigator, Rita Shridharani, Dr. Shridharani, Chattanooga-Hamilton County Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-Lantus
Record Dates: First submitted 2015-09-09; First posted 2015-09-14 (Estimated); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Mellitus, Type 1; Diabetic Ketoacidosis
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Ketoacidosis | interventions — Insulin Glargine; Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Placebo Comparator): The control group will receive all traditional methods of treatment for DKA including iv insulin, correction of fluid loss, and electrolyte correction, including a placebo subcutaneous injection.
  Interventions: Drug: IV insulin; Other: Electrolyte Correction; Other: Correction of Fluid Loss
- Treatment Group (Experimental): The study group will receive the same treatment including iv insulin, correction of fluid loss, and electrolyte correction, but will be supplemented with a subcutaneous glargine injection.
  Interventions: Drug: Glargine; Drug: IV insulin; Other: Electrolyte Correction; Other: Correction of Fluid Loss

INTERVENTIONS:
Drug: Glargine — The control group will receive all traditional methods of treatment for DKA, including a placebo subcutaneous injection. The study group will receive the same treatment, but will be supplemented with a subcutaneous glargine injection.
  Other Names: Lantus
  Arms: Treatment Group
Drug: IV insulin — The intravenous infusion of insulin at a weight-based fixed rate until ketosis has subsided.
Other: Electrolyte Correction — If the potassium level is greater than 6 mEq/L, do not administer potassium supplement. If the potassium level is 4.5-6 mEq/L, administer 10 mEq/h of potassium chloride. If the potassium level is 3-4.5 mEq/L, administer 20 mEq/h of potassium chloride.
Other: Correction of Fluid Loss — Initial correction of fluid loss is either by isotonic sodium chloride solution or by lactated Ringer solution. The recommended schedule for restoring fluids is as follows:
  * Administer 1-3 L during the first hour.
  * Administer 1 L during the second hour.
  * Administer 1 L during the following 2 hours
  * Administer 1 L every 4 hours, depending on the degree of dehydration and central venous pressure readings

SUMMARY:
The management goals of diabetic ketoacidosis (DKA) in the pediatric type 1 diabetes (T1DM) population are fluid and electrolyte repletion, insulin administration, and correction of acidosis in order to stabilize the patient. Traditionally, a rapid-acting insulin IV infusion is begun immediately and continued until the acidosis is corrected and hyperglycemia normalized. Once the acidosis is corrected, patients are able to be transitioned to a subcutaneous insulin regimen.

The role that a subcutaneous long-acting insulin such as glargine has in the acute treatment of DKA has not been extensively studied. While giving glargine during the treatment of DKA is becoming more common place, few studies have examined the potential risks and benefits of its use. This study will investigate the effects of early administration of glargine during DKA in patients with newly diagnosed TIDM.

The design of this study is a prospective, double-blind study of children ages 2-21 who are admitted to the hospital in DKA with a diagnosis of T1DM. The control group will receive all traditional methods of treatment for DKA, including a placebo subcutaneous injection. The study group will receive the same treatment, but will be supplemented with a subcutaneous glargine injection.

ELIGIBILITY:
Inclusion Criteria:

* T1DM
* Hyperglycemia >200 mg/dl
* Bicarbonate ≤ 15 mmol/L
* pH < 7.3
* Ketonemia
* Ketonuria
* Glucosuria
* Admission to PICU (Pediatric Intensive Care Unit)
* Ages 1-21 years

Exclusion Criteria:

* Patients who received glargine within the last 24 hours
* Patients with sepsis

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2015-11; Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Blood glucose | Within 3 hrs of arrival

SECONDARY OUTCOMES:
Blood glucose | 4 hours after intervention initiation
  checking for changes in levels after intervention initiation
blood pH | within 3 hours of arrival
blood pH | 4 hours after intervention initiation
  checking for changes in levels after intervention initiation
blood bicarbonate level | Within 3 hrs of arrival
blood bicarbonate level | 4 hours after intervention initiation
  checking for changes in levels after intervention initiation
Urinalysis for levels of ketones & glucosuria | Within 3 hrs of arrival
Urinalysis for levels of ketones & glucosuria | 4 hours after intervention initiation
  checking for changes in levels after intervention initiation

OTHER OUTCOMES:
Length of PICU Stay | 1-2 days
Length of Hospital Stay | 1-5 days
Hypoglycemic events | length of hospital stay, an expected average of 3 days
  Hypoglycemia is defined as blood glucose less than 70 mg/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Shridharani, MD, Principal Investigator — UTCOMC/ Children's at Erlanger
Locations (1):
- Children's @ Erlanger, Chattanooga, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Levitsky LL et al. Epidemiology, presentation, and diagnosis of type 1 diabetes mellitus in children and adolescents. In: UpToDate, Wolfsdorf J (Ed), UpToDate, Waltham, MA. (Accessed on November 3, 2014.)
- [Background] Jeha GS, Haymond Mw. Treatment and complications of diabetic ketoacidosis in children. In: UpToDate, Waltham MA. (Accessed on November 4, 2014.)
- [Background] Urakami T, Naito Y, Seino Y. Insulin glargine in pediatric patients with type 1 diabetes in Japan. Pediatr Int. 2014 Dec;56(6):822-828. doi: 10.1111/ped.12379. Epub 2014 Sep 16. PMID 24840321
- [Background] Shankar V, Haque A, Churchwell KB, Russell W. Insulin glargine supplementation during early management phase of diabetic ketoacidosis in children. Intensive Care Med. 2007 Jul;33(7):1173-1178. doi: 10.1007/s00134-007-0674-3. Epub 2007 May 17. PMID 17508198
- [Background] Hsia E, Seggelke S, Gibbs J, Hawkins RM, Cohlmia E, Rasouli N, Wang C, Kam I, Draznin B. Subcutaneous administration of glargine to diabetic patients receiving insulin infusion prevents rebound hyperglycemia. J Clin Endocrinol Metab. 2012 Sep;97(9):3132-7. doi: 10.1210/jc.2012-1244. Epub 2012 Jun 8. PMID 22685233
- [Background] 6Lexicomp online